CLINICAL TRIAL: NCT07347548
Title: An Open-label, Single-center, 4-week Phase I Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of Multiple Doses of GRT6019 in Healthy Male Participants
Brief Title: A Trial to Investigate the Safety and Pharmacokinetics of GRT6019 in Healthy Male Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HP6019-07
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Intervention Model Description: Cohorts 1 and 2 will be dosed in parallel, followed by Cohort 3 sequentially
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 4 weeks dosing with GRT6019 once a day [QD]
  Interventions: Drug: GRT6019
- Cohort 2 (Experimental): 4 weeks dosing with GRT6019 once a day [QD]
  Interventions: Drug: GRT6019
- Cohort 3 (Experimental): 4 weeks dosing with GRT6019 once a day [QD]
  Interventions: Drug: GRT6019

INTERVENTIONS:
Drug: GRT6019 — Multiple dose (MD)

SUMMARY:
The purpose of this trial is to assess the safety, tolerability, and PK of 3 doses of GRT6019 in healthy male participants.

This Phase I trial will be a multiple dose trial in healthy male participants with administration of GRT6019 in 3 cohorts.

For each participant, the trial consists of a Screening Period of up to 28 days, a 4 week Treatment Period (including a 2-week clinic stay and 2 weeks in an outpatient setting), and a 5 week Follow-up Period.

DETAILED DESCRIPTION:
There are 8 participants planned per cohort to ensure sufficient sample size for a reliable estimate of PK parameters.

ELIGIBILITY:
Main Inclusion Criteria:

1. Participant must be male, 18 to 55 years of age (inclusive) at the time of signing the informed consent form and affiliated to the social security system.
2. Participant must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
3. Participant must sign the informed consent form before any trial-related assessments.
4. The participant is in good health as determined by the medical history, physical examination, 12-lead ECG, vital signs (heart rate, respiratory rate, systolic and diastolic blood pressure [BP]), body temperature, and clinical laboratory parameters (clinical chemistry, hematology, coagulation, and urinalysis) without clinically relevant (per investigator judgement) deviations from reference ranges unless further specified in the exclusion criteria. The population of this clinical trial is healthy volunteer participants.

Main Exclusion Criteria:

1. Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, comparator, rescue medication, or any ingredients therein, or may affect the interpretation of the results, or may render the participant at high risk from treatment complications/ participation in the study unsafe
2. Major surgical procedure, within 3 months prior to ICF signing, or anticipation of need for a major surgical procedure during the trial
3. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, or immunological disorder(s)
4. Regularly uses any medication, including herbal remedies or over-the-counter medication within 2 weeks before screening into this trial and anticipated use during the trial
5. Concurrent enrollment in another clinical trial, unless it is an observational (non interventional) clinical trial or during the follow-up period of an interventional trial
6. Recent participation in another clinical trial with an IMP administered within 30 days before Day 1 or within 5 times the elimination half-life of the IMP, whichever is longer

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Through study completion, an average of 4 Weeks
  Assessment of safety and tolerability of GRT6019 following 4 weeks of treatment
Number of participants with Serious Adverse Events (SAEs) | Through study completion, an average of 4 Weeks
  Assessment of safety and tolerability of GRT6019 following 4 weeks of treatment
Number of participants with AEs leading to discontinuation | Through study completion, an average of 4 Weeks
  Assessment of safety and tolerability of GRT6019 following 4 weeks of treatment
Number of participants with AEs related to investigational medicinal product [IMP] | Through study completion, an average of 4 Weeks
  Assessment of safety and tolerability of GRT6019 following 4 weeks of treatment

SECONDARY OUTCOMES:
Area under the concentration-time curve over the dosing interval (AUCtau) | Following the first dose (Day 1), then at Day 14, and after the last dose (Day 28)
  Assessment of the pharmacokinetics (PK) of GRT6019 following 4 weeks of treatment, including dose proportionality assessment and investigation of steady state attainment
Maximum observed concentration (Cmax) | Following the first dose (Day 1), then at Day 14, and after the last dose (Day 28)
  Assessment of the pharmacokinetics (PK) of GRT6019 following 4 weeks of treatment, including dose proportionality assessment and investigation of steady state attainment

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial Clinical Pharmacology Unit, Rennes, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Clinical trial transparency at Grünenthal — https://www.grunenthal.com/en/science/clinical-trials